CLINICAL TRIAL: NCT03707782
Title: Mechanisms of Immune Deficiency
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Colorado, Denver (Other)
Collaborators: Colorado Clinical & Translational Sciences Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 18-0337
Record Dates: First submitted 2018-10-12; First posted 2018-10-16 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-04

CONDITIONS: Immune Deficiency
MeSH Terms: conditions — Immunologic Deficiency Syndromes

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood lymphocytes, serum and plasma other tissue if availale
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals with immune deficiencies: aged 18 years or older and have an immune deficiency
- Family members: aged 18 years or older and are related to a person who has an immune deficiency

SUMMARY:
1. The purpose of this study is to learn more about the changes in genes, cells and proteins that cause immune deficiency diseases.
2. The early stages of the study will focus on two groups of patients:

   1. members of families in which several persons have symptoms or medical histories that suggest immune deficiency.
   2. Patients who have received treatments with medications or drugs that affect functions of the immune system (secondary immune deficiencies).

It is hoped that studies will provide guidelines for extension of the research to other patient groups. Up to 200 patients and family members will be invited to participate.

DETAILED DESCRIPTION:
The experiments that are proposed in this portion of the study are intended to:

1. characterize the significance of the variant form of EZH2 identified in this family. They will characterize the degree of methylation of lysine 27 of histone H3 in subjects with the variant and members of the same family who have the wild type gene. The functional methyltransferase activity of the variant and wild type genes will be measured.
2. characterize the current status of B-cell maturation and function in subjects with either the variant gene and the wild type gene.
3. characterize B-cell function (antibody production) and the quality of antibody produced after immunizations in subjects with the wild type gene or the variant gene.

ELIGIBILITY:
Inclusion Criteria:

1. Immunodeficiency disease; or
2. family member of individual with immunodeficiency disease

Exclusion Criteria:

1. Persons with immune deficiencies that are secondary to other diseases such as malignancies.
2. Persons who do not have immune deficiencies, persons who are not meet eligibility criteria

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals aged 18 years or older and have an immune deficiency or are related to a person who has an immune deficiency.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-20 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Measurement of Serum immune globulin | each year for up to 20 years
  The clinical definition of "hypogamma-globulinemia is values that are 2 SD below the mean value for the testing laboratory. For this study values that are below the lower limit of abnormal will be scored as abnormal. Chi-square analysis or Fisher's exact test will compare values between subjects with the wild type gene and the variant gene.
Antibody responses | 4 weeks
  A four-fold difference or a post-immunization titer of ≥1.3 µg/ml is scored as a true antibody response. Antibody titers and avidity indices are transformed to log2 and evaluated using the Student's T-test.
Measurement of NK cell function | one time
  Spearman correlation will be used to compare the relationship between expression of CD207a by NK cells that are activated with K562 cells or NK cells that are activated with PMA/iono.
DNA sequencing | one time
  When indicated, whole exome or whole genome sequencing will be done to identify genetic basis (if any) of the immune deficiency
measurement of cellular components of the immune system | each year for up to 20 years
  Flow cytometry will be used to identify numbers of cells of various types (e.g.,subpopulations of B-cells and T-cells) to evaluate changes in various cell populations over time. This is especially important for studies of family members who carry disease-causing or disease-associated genes but are clinically health at the time of the first study
health outcome measurements | each year for up to 20 years
  The SF-36 form will be used serially to identify changes in health over time
Measurement of avidity | each year for up to 20 years
  avidity indices are transformed to log2 and evaluated using the Student's T-test

CONTACTS AND LOCATIONS:
Overall Officials: Charles Kirkpatrick, Principal Investigator — University of Colorado, Denver
Locations (1):
- UColorado, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bonilla FA, Khan DA, Ballas ZK, Chinen J, Frank MM, Hsu JT, Keller M, Kobrynski LJ, Komarow HD, Mazer B, Nelson RP Jr, Orange JS, Routes JM, Shearer WT, Sorensen RU, Verbsky JW, Bernstein DI, Blessing-Moore J, Lang D, Nicklas RA, Oppenheimer J, Portnoy JM, Randolph CR, Schuller D, Spector SL, Tilles S, Wallace D; Joint Task Force on Practice Parameters, representing the American Academy of Allergy, Asthma & Immunology; the American College of Allergy, Asthma & Immunology; and the Joint Council of Allergy, Asthma & Immunology. Practice parameter for the diagnosis and management of primary immunodeficiency. J Allergy Clin Immunol. 2015 Nov;136(5):1186-205.e1-78. doi: 10.1016/j.jaci.2015.04.049. Epub 2015 Sep 12. PMID 26371839
- [Background] O'Meara MM, Simon JA. Inner workings and regulatory inputs that control Polycomb repressive complex 2. Chromosoma. 2012 Jun;121(3):221-34. doi: 10.1007/s00412-012-0361-1. Epub 2012 Feb 19. PMID 22349693
- [Background] Su IH, Basavaraj A, Krutchinsky AN, Hobert O, Ullrich A, Chait BT, Tarakhovsky A. Ezh2 controls B cell development through histone H3 methylation and Igh rearrangement. Nat Immunol. 2003 Feb;4(2):124-31. doi: 10.1038/ni876. Epub 2002 Dec 23. PMID 12496962
- [Background] Caganova M, Carrisi C, Varano G, Mainoldi F, Zanardi F, Germain PL, George L, Alberghini F, Ferrarini L, Talukder AK, Ponzoni M, Testa G, Nojima T, Doglioni C, Kitamura D, Toellner KM, Su IH, Casola S. Germinal center dysregulation by histone methyltransferase EZH2 promotes lymphomagenesis. J Clin Invest. 2013 Dec;123(12):5009-22. doi: 10.1172/JCI70626. Epub 2013 Nov 8. PMID 24200695
- [Background] Bodor C, Grossmann V, Popov N, Okosun J, O'Riain C, Tan K, Marzec J, Araf S, Wang J, Lee AM, Clear A, Montoto S, Matthews J, Iqbal S, Rajnai H, Rosenwald A, Ott G, Campo E, Rimsza LM, Smeland EB, Chan WC, Braziel RM, Staudt LM, Wright G, Lister TA, Elemento O, Hills R, Gribben JG, Chelala C, Matolcsy A, Kohlmann A, Haferlach T, Gascoyne RD, Fitzgibbon J. EZH2 mutations are frequent and represent an early event in follicular lymphoma. Blood. 2013 Oct 31;122(18):3165-8. doi: 10.1182/blood-2013-04-496893. Epub 2013 Sep 19. PMID 24052547